CLINICAL TRIAL: NCT02270827
Title: A Pilot Study Into Health Pre and Post Treatment With Intravenous Aminophylline and Hydrocortisone in Severe Asthmatics
Acronym: SARAH
Status: Terminated | Type: Observational
Why Stopped: Study was set up by an MSc student who left her post.
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2013AT001B
Record Dates: First submitted 2014-10-06; First posted 2014-10-21 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Aminophylline; Hydrocortisone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aminophylline — intravenous medication
Drug: Hydrocortisone — Intravenous medication

SUMMARY:
This study focuses on severe asthmatics and their asthma symptoms. 40% of asthma patients continue to experience symptoms and up to 5% of these have difficult-to-control asthma despite continually improving treatments. Severe asthmatics experience clinically-significant worse health-related quality of life than those than those with less severe asthma. Poorer health-related quality of life can be as a consequence of frequent, severe symptoms, which prevent the patient from continuing a normal, active lifestyle. The Royal Brompton Hospital uses the treatment regimen of intravenous (IV) Aminophylline and IV Hydrocortisone which appears to improve symptoms and reduce exacerbations. At present there is anecdotal evidence to support these assumptions. The objective of this study is to determine whether there is any objective evidence of improvement, in particular looking at lung function, symptoms and cardiovascular function.

DETAILED DESCRIPTION:
The participant will be involved in this project for approximately 3 - 4 weeks, depending on how long they usually come into hospital for, for clinical treatment. For 1 week they will wear a physical activity monitor before the first course of Aminophylline and Hydrocortisone, during the treatment, and for 1 more week post treatment. This monitor records how active the participants are and is a small monitor worn on the upper arm.

Both study visits will happen while the patients are already in hospital, on admission and on discharge and will take approximately 2-3 hours to complete.

Both study visits include:

• 3 types of breathing tests: Impulse oscillometry in the asthma laboratory, which means they will breath through a mouth piece in and out at a comfortable, steady rate.

Exhaled nitric oxide which measures gas produced by cells in the lungs. This is a comfortable, steady blow into a handheld machine.

Spirometry which involves filling the lungs and blowing out hard into a machine.

* A blood test - Full Blood Count (FBC) including eosinophils, glucose, fibrinogen, C-Reactive Protein (CRP), total Immunoglobulin-E (IgE), citrate coagulation and platelet aggregation.
* 3 short questionnaires which ask about symptoms, control of asthma, and how the patient feels asthma affects them.
* A 6 Minute Walk Test which involves walking up and down a ward corridor for 6 minutes to see distance covered in 6 minutes.
* Cardiovascular test:

Arterial stiffness which is a series of blood pressures on the leg, arm and neck.

Some of these tests will be performed as part of their usual hospital care. These include blood test, 6 Minute Walk Test, and spirometry.

Blood samples will be done routinely as part of normal care. Blood will only be collected if they do not have a clinical blood test before the administration of IV Aminophylline and IV Hydrocortisone and after the final dose. The clinical trial is observing patients on a clinical treatment. All decisions regarding the treatment dose and duration will be made by the clinical team. All samples will go to the standard accredited hospital routine laboratory on the trial site. No samples will be stored, moved off site or leave the UK.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Diagnosis of severe asthma
3. Confirmed therapy adherence via serum Prednisolone and cortisol levels

Exclusion Criteria:

1. Mild and moderate asthma
2. Community acquired pneumonia
3. Acute porphyria
4. Pregnant and breast feeding women
5. Patients hypersensitive to ethylenediamine or allergic to the theophyllines, caffeine and/or theorbromine.
6. Patient with known hypersensitivity to components and in systemic fungal infection
7. Patients that are being administered live attenuated vaccines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe Asthmatic Adults
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To measure a significant improvement in lung function in severe asthmatic patients after receiving a course of IV Aminophylline and IV Hydrocortisone | Day 0 and Day 7 (+/- 3 days)
  Lung function will be measured via spirometry (large airways) and impulse oscillometry (small airways) before and after treatment

SECONDARY OUTCOMES:
To measure a significant improvement in symptoms in severe asthmatic patients after receiving a course of IV Aminophylline and IV Hydrocortisone | Day 0 and Day 7 (+/- 3 days)
  This will be measured by looking at symptoms via 2 questionnaires, ACQ-7, Dyspnoea-12, before and after treatment
To measure a significant improvement in quality of life in severe asthmatic patients after receiving a course of IV Aminophylline and IV Hydrocortisone | Day 0 and Day 7 (+/- 3 days)
  This will be measured by giving each patient the EuroQOL questionnaire before and after treatment
To measure a significant improvement in exercise tolerance in severe asthmatic patients after receiving a course of IV Aminophylline and IV Hydrocortisone | Day 0 and Day 7 (+/- 3 days)
  This will be measured by asking each patient to perform a 6 Minute Walk Test before and after treatment
To measure a significant cardiovascular change in severe asthmatic patients after receiving a course of IV Aminophylline and IV Hydrocortisone | Day 0 and Day 7 (+/- 3 days)
  This will be measured by performing Arterial Stiffness on each patient which involves measuring a series of blood pressures on the carotid, femoral and brachial arteries before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Menzies-Gow, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom